CLINICAL TRIAL: NCT06384885
Title: Ultrasound Investigation Into Swimming Induced Pulmonary Edema in Open Water Swimming Athletes
Acronym: SIPE
Status: Recruiting | Type: Observational
Sponsor: Rocky Vista University, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-079
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Swimming Induced Pulmonary Edema
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Triathletes/Open water swimmers: Triathletes and open water swimmers in events at Boulder Ironman, St George Ironman and Without limits swim events
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Lung ultrasound

SUMMARY:
Swimming-induced pulmonary edema (SIPE) is a potentially life-threatening condition that can affect swimmers of all abilities. The pathophysiology is not well understood and early identification strategies are not established. Handheld ultrasound is a validated tool for the identification of pulmonary edema and is not well-studied in this population. Understanding the incidence of signs of pulmonary edema and its usefulness as a sign of early pulmonary edema would be beneficial This study evaluates triathletes and open water swimmers at endurance events. A validated protocol for lung ultrasound is used to identify the signs of pulmonary edema. The findings will be analyzed for differences in experience level, type of athlete, gender, age, and environmental factors. The findings may then be used in the future to aid in the early identification and treatment of athletes and military personnel in similar situations to decrease morbidity and mortality.

DETAILED DESCRIPTION:
This research project aims to advance the understanding of the signs of pulmonary edema by evaluating both symptomatic and asymptomatic individuals at triathlons and open water swim events. Ultrasound is being used here as it is a validated tool for the assessment of pulmonary edema and pleural effusion and is highly portable and cost-effective, improving access to imaging in austere and limited-resource medical environments.

Swimming-induced pulmonary edema lacks an abundance of evidence identifying its pathophysiology, as well as information regarding the normal progression of signs and symptoms. Unfortunately, while there are some protocols for identifying patients with symptoms, many times these are too late and symptoms are advanced. Improving the identification of early signs of SIPE may lead to better outcomes, more timely intervention, and an improved understanding of the pathophysiology of the disease.

Use of a high-quality handheld ultrasound to evaluate open-water swimmers for signs of pulmonary edema will contribute to the field in several ways. First, improving knowledge of the signs in both symptomatic and asymptomatic individuals is beneficial to the identification and early treatment of patients. Secondly, utilizing portable imaging technology for novel applications improves utility and may increase access to medical resources in resource-poor environments. Third, by validating this protocol for the evaluation of SIPE, medical professionals who attend to patients who may experience SIPE have improved diagnostic capability to intervene earlier. Literature shows a higher incidence of SIPE in military training recruits, such as Navy Seals, and open-water swimming athletes, both of whom operate in austere and resource-limited environments, and would benefit from improved early diagnostic tools to identify pathology.

Our specific aims are to utilize ultrasound and the BLUE protocol (described below), and acquisition of vital signs, and health history in the medical tent with patients and with a control group of race finishers to identify normal anatomy or pathology. We will compare findings in areas of previous experience, level of fitness, gender, age, wetsuit status, and environmental factors. We will run a statistical analysis to compare our findings and account for the day's environmental factors, race type, history, and physical exam findings.

Swimming Induced Pulmonary Edema (SIPE), is a poorly understood respiratory pathology that can affect individuals without underlying health conditions and can be potentially life-threatening. (Spencer, 2018). SIPE is an immersion pulmonary edema presenting with dyspnea, chest pain, cough, hemoptysis, frothy sputum production, and may result in death. (miller 2011) (Grunig 2017) ( Smart, 2014) (Department of the Navy, 2023). The pathophysiological mechanisms of SIPE are not fully understood but may involve the redistribution of blood centrally during cold water immersion, resulting in elevated pressure in the right-sided intravascular system and a concurrent increase in afterload (Wester 2009). Some individuals with a history of SIPE tend to have increased Mean Pulmonary Artery Pressure (MPAP) and Pulmonary Artery Wedge Pressure (PAWP)with a reduction in these pressures and SIPE incidence after a 50 mg oral dose of sildenafil. Understanding the pathophysiology of SIPE considers its multifaceted causes consisting of environmental, genetic, and predisposing risk factors. (Moon 2016).

In triathletes, the prevalence of SIPE has been reported as high as 1.4% (Miller, 2010), and reports of SIPE symptoms range from 1.8-6.0% in combat swimmer trainees during a 2.4-3.6 km open ocean swim (Shupak et al, 2000),. Unlike military swimmers or competitive swimmers, triathlete athletes may not have formal training, coaching, and competition experience in swimming, including open water swim which brings about the added challenges of previous training, environmental conditions, navigation, and absence of lane markers. The varied levels of experience in stroke quality, timing, breathing timing, or subsequent physical activity (bike and run) and the incidence of SIPE have not been studied and are areas for further investigation.

Ultrasound has proven methodology to diagnose pulmonary edema and has proven to be effective in diagnosing pulmonary edema post open water swim, including in patients who had no prior history of pulmonary edema, preexisting conditions, or inciting factors other than open water swim, suggesting that the pathology was a form of immersion pulmonary edema induced by swimming. (parasuraman et al 2016) (Hardstedt et al 2021). An algorithm suggested for SIPE diagnosis uses ultrasound to validate symptomologic criteria, including SPO2, lung sounds, and sputum production. However, lung ultrasound has not been utilized to investigate possible signs of pulmonary edema in asymptomatic patients who present following an open-water swim or immersion event. (hardstedt et al, 2020). Early identification of signs of SIPE is highly beneficial in preventing morbidity and mortality in military and athletes. Long-term benefits from this study include using this data for future events to develop protocols using ultrasound to aid in early detection and treatment ultimately reducing morbidity and mortality.

Our team's previous work in this field will help the current research. Our faculty PI recently authored part of a book chapter describing ultrasound findings in SIPE. All members of the research team have previous experience volunteering in medical tents at endurance events. The faculty PI has been the medical director for several endurance events and helped develop and use specific protocols for commonly seen emergent medical issues at these events. Our researchers have various POCUS and ARDMS ultrasound certifications. Additionally, both researchers are involved in an ultrasound scholar program that runs longitudinally with their coursework and provides rigorous training and hands-on experience in ultrasound diagnostics that provide a relevant foundation to the current research. One team member has experience in the development and delivery of an ultrasound curriculum to first-year medical students and high school learners focused on a comprehensive understanding of ultrasound use with an additional emphasis on emergent events and sports-related evaluations. The other lead researcher on our team has experience coordinating austere medical care, for private organizations providing ICU and ED level care to races, mass gatherings, concerts, and disasters, as well as coordinating resource medical limited care for government agencies. He has been awarded multiple grants to conduct research in the instruction and utilization of ultrasound in remote and austere environments to improve the early diagnostic capability of physicians as well as other medical providers.

Our study will utilize a prospective observational cohort study to investigate the incidence and risks associated with SIPE in athletes after the swimming leg of an IronMan race or open water swimming event. We will additionally be present at other races, working collaboratively with the medical staff that organizes the care at these races. The company is called Rapid Response Paramedic Services. Study participants will be stable, non-emergent athletes recruited from multiple medical tents at the event. Upon initial medical treatment, participants will complete a survey and undergo a physical examination to determine their symptomatology related to SIPE, and further categorized as either asymptomatic or symptomatic using the criteria outlined below.

The study will assess the burden of SIPE in asymptomatic individuals following the swimming leg of the race using an algorithm that incorporates lung ultrasound as the major diagnostic methodology. POCUS of the lung will be performed utilizing the Bedside Lung Ultrasound Examination (BLUE protocol) as a guide. Confirmation of pulmonary edema will be determined by ultrasound and we will associate these findings with symptoms, or lack thereof experienced by the athletes. Additionally, our data will be documented sequentially to determine the timing of symptoms and ultrasound findings in relation to the completion of the swimming leg of the race and its association with other legs of the race (running/cycling). The study will also include scanning of symptomatic individuals (if non-emergent and stable) for comparative analysis but will focus primarily

Further Breakdown of Inclusion into Symptomatic and Asymptomatic Groups:

Symptomatic Group:

Participants who self-report symptoms of Swimming-Induced Pulmonary Edema (SIPE) such as cough, dyspnea, increased sputum, hemoptysis, or a combination thereof.

Lung auscultation findings that include crackles, rhonchi, or other abnormalities.

Participants with SPO2 levels below 95% and/or abnormal lung sounds on auscultation.

Asymptomatic Group:

Participants who do not report any symptoms of SIPE. Participants with SPO2 levels of 95% or above and normal lung sounds on auscultation.

Equipment List:

Ultrasound:

1. Butterfly IQ + Ultrasound Device
2. Medsong Ltd Portable Ultrasound
3. GE VSCAN CL portable ultrasound
4. Ultrasound Gel
5. Probe Wipes
6. iPad

Medical Equipment:

1. Stethoscopes
2. Pulse Oximeters
3. Blood Pressure Monitors
4. Cardiac monitor
5. Thermometer

Survey Equipment:

1. Tablets/Laptops with survey software
2. Stopwatch

PPE + Misc:

1. Gloves + Hand Sanitizer 2. Towels 3. Tape, Markers, Pens, Storage Study population and settings

1. The Study population: Will consist of previously healthy open water swimming athletes that are dropping from the race after (OR DURING) the swimming leg; Or have finished the race and are seeking medical attention post race.
2. The study setting: Participants will be recruited from the medical tents at the IronMan or open water swimming race. Ultrasound scanning and data collection will take place at the same location. The location will differ depending on the event, but all events will be in conjunction with the company Rapid Response Paramedic Services.

This initial prospective cohort study will be conducted during the IRONMAN 70.3 Boulder race in Boulder, Colorado, on June 8, 2024, and potentially at a subsequent race in Utah (specific date to be confirmed). Eligible participants must be 18 years of age or older, have completed the swimming leg of the race, and either have dropped out or completed the race, reporting to the medical tent with a stable presentation (refer to the exclusion criteria above).

Inclusion and Exclusion Criteria

Inclusion Criteria:

* Participants must be Athletes competing in the event
* Must have engaged in a portion of the swimming leg of the race

Exclusion Criteria:

* Any acutely decompensating patient who requires focused medical care and evacuation as determined by race physicians
* Patients who are pregnant
* Patients less than 18 years of age

Validated SIPE Diagnostic Criteria

"Algorithm for SIPE diagnosis in patients with acute onset of cough and/or dyspnea during swimming in open water. The algorithm is based on peripheral oxygen saturation (SpO2) and crackles on lung auscultation, with excessive sputum and/or hemoptysis supporting the diagnosis. Patients with findings of crackles and SpO2 ≤95% could be diagnosed with SIPE based on clinical evaluation. For patients with findings of crackles or SpO2 ≤95%, lung ultrasound (LUS) is suggested for differential diagnosis if available." Previously published by Hårdstedt et al, CHEST 2020 and utilized in Hardstedt et al, in CHEST 2021.

Lung Ultrasound Protocol and Examination Lung ultrasound will be performed on every individual included in the study. Our lung ultrasound exam is derived from the Bedside Lung Ultrasound Examination developed and published in the Lung Ultrasound in the Criticall Ill (Lichtenstein, 2014). Our exam will establish positive lung sliding and determine if a B-Profile is present in the individuals. The BLUE protocol establishes a 97% sensitivity, 95% specificity, 87% positive predictive value, and 99% negative predictive value in determining acute hemodynamic pulmonary edema in patients who present with a B-profile. (Lichtenstein, 2014). A B-profile indicating bilateral pulmonary edema included 3 or more b lines in all 4 BLUE points, however we also include 3 or more B lines unilaterally in 2 BLUE points, indicating unilateral pulmonary edema.

Figure: BLUE Protocol (Bedside Lung Ultrasound Examination) from which our modifications were made from. We aimed to identify 3 or more B-lines on lung ultrasound to state with >90% sensitivity that pulmonary edema was present.

Figure: Scan locations using a convex probe on each athlete. Areas of investigation and the BLUE-points. Two hands placed this way (size equivalent to the patient's hands, upper hand touching the clavicle, thumbs excluded) correspond to the location of the lung, and allow three standardized points to be defined. The upper-BLUE-point is at the middle of the upper hand. The lower-BLUE-point is at the middle of the lower palm. The PLAPS-point is defined by the intersection of: a horizontal line at the level of the lower BLUE-point; a vertical line at the posterior axillary line. Small probes, such as this Japanese microconvex one (1992), allow positioning posterior to this line as far as possible in supine patients, providing more sensitive detection of posterolateral alveolar or pleural syndromes (PLAPS). The diaphragm is usually at the lower end of the lower hand. Extract from "Whole body ultrasonography in the critically ill" (2010 Ed, Chapter 14), (Lichtenstein, 2011)

Both the physical examinations and the ultrasound examinations will be conducted by researchers, which include medical students. Each physical examination and ultrasound study will be monitored by a physician or certified healthcare professional from Rapid Response Paramedic Services, they will all be in the same room, and images saved from the ultrasound exam will be examined by the physician for diagnosis. In the event of a mistake or error in the physical exam or diagnosis, the licensed healthcare professional will intervene to correct the error. Limitations in this study include the remote environment. If an individual decompensates they will be directed to the care of the Rapid Response Paramedic Services medical team and may be lost to followup. Additionally, due to the high-intensity nature of athletic events, it is possible that responses to our health history questionnaire may be brief and omit some information that might not be omitted in a traditional healthcare setting, to compensate for this we have developed a healthcare questionnaire that is standardized to be used with all patients. Finally, we may have a selection bias due to conducting the study in the medical tent, we may not receive as many asymptomatic individuals as symptomatic individuals seeking additional care, to compensate for this we will add additional advertising outside the tented areas, requesting any individual interested in supporting athlete medial research join the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Participants must be Athletes competing in the event
* Must have engaged in a portion of the swimming leg of the race

Exclusion Criteria:

* - Any acutely decompensating patient who requires focused medical care and evacuation as determined by race physicians
* Patients who are pregnant
* Patients less than 18 years of age
* Athletes who did not participate in the swim portion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Triathletes and open water swimmers at participating races.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasound | at triathlon- immediately after race
  Evaluate for significant amount of B lines

CONTACTS AND LOCATIONS:
Locations (1):
- Rocky Vista University, Parker, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Make available to other researchers of open water events through academic sports medicine channels
Supporting Information: Study Protocol
Time Frame: starting 2025 and ongoing
Access Criteria: They will need to contact us to share data

REFERENCES:
- [Background] Morgan WJ, Taussig LM. The chronic bronchitis complex in children. Pediatr Clin North Am. 1984 Aug;31(4):851-64. doi: 10.1016/s0031-3955(16)34649-1. PMID 6146959
- [Background] Toker C. Observations on the ultrastructure of a mammary ductule. J Ultrastruct Res. 1967 Nov;21(1):9-25. doi: 10.1016/s0022-5320(67)80003-0. No abstract available. PMID 5583207
- [Background] Peirce EC 2nd. A comparison of the Lande-Edwards, the Peirce, and the General Electric-Peirce membrane lungs. Trans Am Soc Artif Intern Organs. 1970;16:358-64. No abstract available. PMID 5454185
- [Background] Hardstedt M, Seiler C, Kristiansson L, Lundeqvist D, Klingberg C, Braman Eriksson A. Swimming-Induced Pulmonary Edema: Diagnostic Criteria Validated by Lung Ultrasound. Chest. 2020 Oct;158(4):1586-1595. doi: 10.1016/j.chest.2020.04.028. Epub 2020 Apr 28. PMID 32360726
- [Background] Woollard KV. The Quality in Australian Health Care Study. Med J Aust. 1996 Mar 4;164(5):315. doi: 10.5694/j.1326-5377.1996.tb94205.x. No abstract available. PMID 8628172
- [Background] Wester TE, Cherry AD, Pollock NW, Freiberger JJ, Natoli MJ, Schinazi EA, Doar PO, Boso AE, Alford EL, Walker AJ, Uguccioni DM, Kernagis D, Moon RE. Effects of head and body cooling on hemodynamics during immersed prone exercise at 1 ATA. J Appl Physiol (1985). 2009 Feb;106(2):691-700. doi: 10.1152/japplphysiol.91237.2008. Epub 2008 Nov 20. PMID 19023017